CLINICAL TRIAL: NCT04478032
Title: Deep Transcranial Magnetic Stimulation for the Treatment of Treatment Resistance Schizophrenia: a Double-Blind, Randomized Clinical Trial
Brief Title: Deep Transcranial Magnetic Stimulation for the Treatment of Treatment Resistance Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20194Y0037
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-07

CONDITIONS: Deep Transcranial Magnetic Stimulation for the Treatment of Treatment Resistance Schizophrenia
Keywords: Treatment Resistance Schizophrenia; Deep Transcranial Magnetic Stimulation; anterior cingulate cortex; glutamate; H7 coil

STUDY DESIGN:
Intervention Model Description: In this research,we combine a cross-sectional case control study and a randomized controlled study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham stimulation (Sham Comparator): 20 patients will be randomly allocated into this group,they will receive sham stimulation.
  Interventions: Device: deep transcranial magnetic stimulation with H7 coil
- real stimulation dTMS targeting the ACC (Active Comparator): 20 patients will be randomly allocated into this group,they will receive real stimulation.
  Interventions: Device: deep transcranial magnetic stimulation with H7 coil

INTERVENTIONS:
Device: deep transcranial magnetic stimulation with H7 coil — low frequency(1Hz) deep transcranial magnetic stimulation on ACC .Duration:20 days.

SUMMARY:
Based on the hypothesis that low-frequency deep transcranial magnetic stimulation(dTMS) on anterior cingulate cortex （ACC） could down-regulate the glutamate level of ACC and regulate the acc-related functional network in patients with treatment resistance schizophrenia,this research plan to utilise multimodal functional magnetic imaging method(including structural MRI,resting-state functional magnetic resonance imaging and 1H-MRS) to investigate therapeutic efficacy of low-frequency deep transcranial magnetic stimulation on SZ patients symptoms,as well as to elucidate the correlation between treatment effects and glutamate level of ACC

DETAILED DESCRIPTION:
This study includes 20 treatment resistance schizophrenia patients and 20 healthy controls.This study will investigate 1)abnormalities of the glutamate level of ACC in patients with schizophrenia compared to healthy controls by using 1H-MRS technique. 2)potential modulation effects of deep transcranial magnetic stimulation(dTMS) on anterior cingulate cortex function of patients with schizophrenia. 3)the therapeutic efficacy of dTMS on cognitive impairments and other psychotic symptoms of patients with schizophrenia by adopting cognitive function and psychotic symptoms evaluation,as well as to explore the optimal dTMS treatment pattern on cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia who meet the dsm-5 diagnostic criteria
* Aged from 18 to 60
* After 4 weeks of treatment with a sufficient dose of an antipsychotic (equivalent dose of 400 ~ 600 mg/ day chlorpromazine (CPZ)), no clinical improvement was achieved (at least two items in PANSS scale P1,P2,P3,N1,N4,N6,G5 and G9 ≥4 points, or cgi-s ≥4 points)
* Right-handedness, normal hearing, visual acuity or corrected visual acuity
* Written informed consent of the patient and his/her family

Exclusion Criteria:

* Patients who are currently taking clozapine or who have failed to respond to a full course of treatment with clozapine
* Current or past neurological illness,severe physical illness,substance abuse or addiction,alcohol dependence,mental retardation,pregnancy or lactation,extreme agitation, stupor, negative suicide,or those who can not cooperate
* A history of MECT within 6 months,or those with contraindications to MRI,rTMS
* Medically unstable for at least 1 month (PANSS score fluctuation>10%)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-07-05 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale(PANSS) | baseline,24 hours after the dTMS treatment,30 days
  Change from baseline in Positive and Negative Syndrome Scale(PANSS) after dtms treat 30 days
Change from baseline in MATRICS Consensus Cognitive Battery | baseline,24 hours after the rTMS treatment,30 days
  MATRICS Consensus Cognitive Battery

SECONDARY OUTCOMES:
Change of ACC neurogenesis | baseline,24 hours after the dTMS treatment
  Quantify neural stem cells in hippocampal by using H1-MRS
Change in glutamate level | baseline,24 hours after the dTMS treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No